CLINICAL TRIAL: NCT02880475
Title: An Open-label, Randomized, Single-dose, Parallel Group Study to Investigate the Pharmacokinetics of Oxycodone and Naloxone From OXN 5/2.5 and OXN 20/10 in Chinese Patients With Moderate to Severe Chronic Non-malignant Pain
Brief Title: OXN PR Tablet 5/2.5 mg and20/10 mg PK Study in Chinese Moderate to Severe Chronic Non-malignant Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mundipharma (China) Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OXN08-CN-101
Record Dates: First submitted 2016-07-26; First posted 2016-08-26 (Estimated); Results first posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-04

CONDITIONS: Chronic Pain
Keywords: Moderate to severe chronic non-malignant pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OXN prolonged release tablet 5/2.5mg (Experimental): The subjects were randomized to receive a single dose of OXN prolonged release tablet 5/2.5mg for one time.
  Interventions: Drug: OXN PR tablet
- OXN prolonged release tablet 20/10mg (Experimental): The subjects were randomized to receive a single dose of OXN prolonged release tablet 20/10 mg for one time.
  Interventions: Drug: OXN PR tablet

INTERVENTIONS:
Drug: OXN PR tablet — Orally administered OXN PR tablet 5/2.5 mg or OXN PR tablet 20/10 mg
  Other Names: Targin

SUMMARY:
This is an open-label, randomized, single-dose, parallel group study. The objectives of this study are to assess pharmacokinetics of oxycodone and naloxone from oxycodone/naloxone (OXN) prolonged release (PR) tablet 5/2.5 mg (OXN 5/2.5) and 20/10 mg (OXN 20/10) in Chinese patients with moderate to severe chronic non-malignant pain.

DETAILED DESCRIPTION:
It will be conducted to assess the pharmacokinetics of OXN 5/2.5 and OXN 20/10 tablets. Subjects will be allocated to a sequence of two strength group in accordance with a random allocation schedule (RAS) in a 1:1 ratio.

Subjects will attend a screening visit within 14 days of the first (OXN) dosing day (Day 1).

Eligible subjects will then check into the study unit on the day before OXN dosing (Day -2). Subjects will be administered their OXN dose the next 2 morning (Day 1), following an overnight fast.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Chinese patients with moderate to severe chronic non-malignant pain.
2. Male and female subjects with age range 18 to 65 years (including 18 and 65), body weight ≥ 45kg and BMI range 18 to 30 (including 18 and 30).
3. Patients who should rate their pain (Pain Intensity Scale -"average pain" over the last 24 hours) as ≥4 on 0-10 scale.
4. Patients, who are able to read, understand and sign written informed consent prior to study participation and are willing to follow the protocol requirements.
5. Females of childbearing potential and less than one year post-menopausal must have a negative serum pregnancy test during screening visit and at check-in and be non-lactating. In addition, they must be willing to use adequate and reliable contraception throughout the study. Highly effective methods of birth control are defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as sterilization, implants, injectables, combined oral contraceptives, some IUDs (intrauterine Device, hormonal), sexual abstinence or vasectomised partner.

Exclusion Criteria:

1. Females who are pregnant (positive β-human chorionic gonadotrophin [HCG] test) or lactating.
2. Use of opioid or opioid antagonist-containing medication in the 30 days before the start of the study.
3. Known sensitivity to oxycodone, naloxone, or related compounds.
4. Subjects with clinically unstable respiratory disease, dysfunction of the biliary tract, thyroid disease, adrenal cortical insufficiency, prostatic hypertrophy requiring intervention (medication or surgical) or renal artery stenosis, or any other medical condition, that, in the opinion of the investigator or the sub-investigator, precludes entry into this study.
5. Subject who have a past (within 5 years) history of malignant neoplasm including leukemia and lymphoma.
6. The electrocardiogram examination results are abnormal, in the opinion of the investigator or the sub-investigator, and are clinical significance.
7. Subjects with abnormal liver function (values exceed the upper limit of normal for AST, ALT or total bilirubin during the Screening Period) or abnormal renal function (values exceed the upper limit of normal for serum creatinine during the Screening Period).
8. Patients with a contraindication to the study medication.
9. Subjects who have a psychiatric disorder such that participation in the study may, in the opinion of the investigator or the sub-investigator, pose an unacceptable risk to the subject.
10. Subjects who have a current or past (within 5 years) history of substance or alcohol abuse, or subjects who give a positive result in drug abuse test during the Screening Period, or subjects who, in the opinion of the investigator or the sub-investigator, have demonstrated addictive or substance abuse behaviors.
11. Subjects with uncontrolled seizures or convulsive disorder.
12. Subjects who will receive any interventional therapy (surgery, paracentesis,etc) for arthritis during the study period.
13. History of or any current conditions that might have interfered with drug absorption, distribution, metabolism or excretion.
14. Any history of frequent nausea or emesis regardless of aetiology.
15. Participation in any clinical drug study during the 3 months preceding the initial dose in this study.
16. Use of any medication including vitamins, herbal and/or mineral supplements during the course of the study, other than Vitamin D, calcium supplements and continued use by females of contraceptive medication or HRT.
17. Consumption of alcoholic beverages within 48 hours before study drug administration, and refusal to abstain from alcohol until at least 48 hours after the last study drug administration.
18. Blood or blood products donated within 90 days prior to study drug administration or anytime during the study, except as required by this protocol.
19. Positive results of urine drug screen(for opioids, barbiturates, amphetamines, cocaine metabolites, methadone, diazepam and cannabinoids), alcohol breath test, hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (Ab), human immunodeficiency virus (HIV) test or qualitative syphilis tests.
20. Patients with moderate to severe hypohemia (HGB<90g/L during the screening).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2015-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria YU, Study Director — Mundipharma (China) Pharmaceutical Co. Ltd
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- OXN Prolonged Release Tablet 5/2.5 mg: The subjects were randomized to receive a single dose of OXN prolonged release tablets 5/2.5mg for one time.
  OXN PR tablet: Orally administered OXN PR tablet 5/2.5 mg
- OXN Prolonged Release Tablet 20/10 mg: The subjects were randomized to receive a single dose of OXN prolonged release tablets 20/10mg for one time.
  OXN PR tablet: Orally administered OXN PR tablet 20/10 mg
Period: Overall Study
Arm/Group | OXN Prolonged Release Tablet 5/2.5 mg | OXN Prolonged Release Tablet 20/10 mg
Started | 13 | 17
Completed | 13 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- OXN PR Tablet 5/2.5 mg; OXN PR Tablet 20/10 mg: The subjects will be randomized to receive either a single dose of OXN prolonged release tablets 5/25mg, 20/10 mg for one time.
  OXN PR tablet: Orally administered OXN PR tablet 5/2.5 mg or OXN PR tablet 20/10 mg
- Total: Total of all reporting groups
Arm/Group | OXN PR Tablet 5/2.5 mg | OXN PR Tablet 20/10 mg | Total
Number analyzed (Participants) | 13 | 17 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 17 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 6 | 9 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 13 | 17 | 30

OUTCOME MEASURES:

1. Primary Outcome: AUC0-48hr of Noroxycodone Plasma Concentration.
Description: AUC0-48hr of Noroxycodone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg will be analyzed.
Time Frame: Pre-dose, 0.5h, 1.0h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 7h, 8h, 10h, 12h, 14h, 24h, 28h, 32h, 36h, and 48h Post Dose blood sampling to determine the PK of oxycodone and metabolites in Chinese patients.
Population: 12 subjects in OXN PR tablet 5/2.5 mg group,12 subjects in OXN PR tablet 20/10 mg group.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | OXN PR Tablet 5/2.5 mg | OXN PR Tablet 20/10 mg
Number analyzed (Participants) | 12 | 12
hr*ng/mL | 81.72 (39.82) | 325.51 (99.47)

2. Primary Outcome: AUC0-t of Noroxycodone Plasma Concentration
Description: AUC0-t of Noroxycodone plasma concentration.Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg will be analyzed .(If the extrapolated area of AUC is larger than 20% of AUCinf, i.e. AUC0-t/AUCinf < 0.8, then the elimination-related PK parameters (AUCinf, T1/2, Lambda_z) will not be adopted and will not be included in any statistical analysis. )
Time Frame: as for outcome 1
Population: 12 subjects in OXN PR tablet 5/2.5 mg group,12 subjects in OXN PR tablet 20/10 mg group.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Groups:
- OXN Prolonged Release Tablet 5/2.5mg: The subjects will be randomized to receive either a single dose of OXN prolonged release tablets 5/2.5mg for one time.
  OXN PR tablet: Orally administered OXN PR tablet 5/2.5 mg or OXN PR tablet 20/10 mg
- OXN Prolonged Release Tablet 20/10mg: The subjects will be randomized to receive either a single dose of OXN prolonged release tablets 20/10 mg for one time.
  OXN PR tablet: Orally administered OXN PR tablet 5/2.5 mg or OXN PR tablet 20/10 mg
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr*ng/mL | 81.25 (40.27) | 325.37 (99.76)

3. Primary Outcome: AUC_%Extrap of Noroxycodone Plasma Concentration
Description: AUC_%Extrap of Noroxycodone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: Pre-dose, 0.5h, 1.0h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 7h, 8h, 10h, 12h, 14h, 24h, 28h, 32h, 36h, and 48h Post Dose blood sampling to determine the PK of oxycodone, naloxone and metabolites in Chinese patients.
Measure: Mean (Standard Deviation); unit: (%)
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
(%) | 2.99 (1.17) | 1.45 (0.67)

4. Primary Outcome: AUCinf of Noroxycodone Plasma Concentration
Description: AUCinf of Noroxycodone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr*ng/mL | 83.74 (41.66) | 330.44 (102.51)

5. Primary Outcome: Cmax of Noroxycodone Plasma Concentration
Description: Cmax of Noroxycodone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
ng/mL | 4.68 (1.53) | 20.69 (3.88)

6. Primary Outcome: Lambda_z of Noroxycodone Plasma Concentration
Description: Lambda_z of Noroxycodone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
1/hr | 0.10 (0.02) | 0.10 (0.01)

7. Primary Outcome: T1/2 of Noroxycodone Plasma Concentration
Description: T1/2 of Noroxycodone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr | 7.42 (1.42) | 7.16 (1.02)

8. Primary Outcome: Tmax of Noroxycodone Plasma Concentration
Description: Tmax of Noroxycodone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Median (Full Range); unit: hr
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr | 4.50 [1.50 to 8.02] | 4.00 [2.50 to 5.02]

9. Primary Outcome: AUC0-48hr of Noroxymorphone Plasma Concentration
Description: AUC0-48hr of Noroxymorphone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr*ng/mL | 14.10 (5.02) | 65.84 (25.50)

10. Primary Outcome: AUC0-t of Noroxymorphone Plasma Concentration
Description: AUC0-t of Noroxymorphone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr*ng/mL | 12.92 (5.21) | 65.65 (25.78)

11. Primary Outcome: AUC_%Extrap of Noroxymorphone Plasma Concentration
Description: AUC_%Extrap of Noroxymorphone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: (%)
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
(%) | 14.89 (11.61) | 4.25 (1.98)

12. Primary Outcome: AUCinf of Noroxymorphone Plasma Concentration
Description: AUCinf of Noroxymorphone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr*ng/mL | 15.76 (4.68) | 68.17 (26.22)

13. Primary Outcome: Cmax of Noroxymorphone Plasma Concentration
Description: Cmax of Noroxymorphone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
ng/mL | 0.75 (0.29) | 3.54 (1.64)

14. Primary Outcome: Lambda_z of Noroxymorphone Plasma Concentration
Description: Lambda_z of Noroxymorphone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
1/hr | 0.08 (0.02) | 0.08 (0.01)

15. Primary Outcome: T1/2 of Noroxymorphone Plasma Concentration
Description: T1/2 of Noroxymorphone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr | 8.55 (1.53) | 9.08 (1.42)

16. Primary Outcome: Tmax of Noroxymorphone Plasma Concentration
Description: Tmax of Noroxymorphone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Median (Full Range); unit: hr
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr | 7.00 [2.00 to 10.00] | 5.00 [2.50 to 7.00]

17. Primary Outcome: AUC0-48hr of Oxycodone Plasma Concentration
Description: AUC0-48hr of Oxycodone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr*ng/mL | 89.48 (34.38) | 272.11 (48.51)

18. Primary Outcome: AUC0-t of Oxycodone Plasma Concentration
Description: AUC0-t of Oxycodone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr*ng/mL | 88.45 (34.55) | 271.21 (48.79)

19. Primary Outcome: AUC_%Extrap of Oxycodone Plasma Concentration
Description: AUC_%Extrap of Oxycodone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: (%)
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
(%) | 1.78 (1.15) | 0.57 (0.21)

20. Primary Outcome: AUCinf of Oxycodone Plasma Concentration
Description: AUCinf of Oxycodone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr*ng/mL | 89.85 (34.72) | 272.71 (48.77)

21. Primary Outcome: Cmax of Oxycodone Plasma Concentration
Description: Cmax of Oxycodone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
ng/mL | 6.69 (1.67) | 24.64 (6.30)

22. Primary Outcome: Lambda_z of Oxycodone Plasma Concentration
Description: Lambda_z of Oxycodone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
1/hr | 0.14 (0.04) | 0.14 (0.02)

23. Primary Outcome: T1/2 of Oxycodone Plasma Concentration
Description: T1/2 of Oxycodone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr | 5.09 (0.96) | 5.03 (0.69)

24. Primary Outcome: Tmax of Oxycodone Plasma Concentration
Description: Tmax of Oxycodone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Median (Full Range); unit: hr
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr | 3.75 [1.02 to 8.00] | 2.00 [0.50 to 5.00]

25. Primary Outcome: AUC0-48hr of Oxymorphone Plasma Concentration
Description: AUC0-48hr of Oxymorphone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr*ng/mL | 3.70 (1.33) | 3.59 (0.97)

26. Primary Outcome: AUC0-t of Oxymorphone Plasma Concentration
Description: AUC0-t of Oxymorphone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr*ng/mL | 0.14 (0.33) | 1.66 (1.21)

27. Primary Outcome: AUC_%Extrap of Oxymorphone Plasma Concentration
Description: AUC_%Extrap of Oxymorphone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: (%)
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
(%) | 82.85 (21.51) | 51.11 (26.70)

28. Primary Outcome: AUCinf of Oxymorphone Plasma Concentration
Description: AUCinf of Oxymorphone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Population: If the extrapolated area of AUC is larger than 20% of AUCinf, i.e. AUC0-t/AUCinf < 0.8, then the elimination-related PK parameters (AUCinf, T1/2, Lambda_z) will not be adopted and will not be included in any statistical analysis.
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 0 | 0

29. Primary Outcome: Cmax of Oxymorphone Plasma Concentration
Description: Cmax of Oxymorphone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
ng/mL | 0.03 (0.06) | 0.30 (0.17)

30. Primary Outcome: Lambda_z of Oxymorphone Plasma Concentration
Description: Lambda_z of Oxymorphone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Population: as for outcome 28
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 0 | 0

31. Primary Outcome: T1/2 of Oxymorphone Plasma Concentration
Description: T1/2 of Oxymorphone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Population: as for outcome 28
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 0 | 0

32. Primary Outcome: Tmax of Oxymorphone Plasma Concentration
Description: Tmax of Oxymorphone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Median (Full Range); unit: hr
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr | 0.75 [0.50 to 1.00] | 1.75 [0.50 to 5.00]

33. Primary Outcome: AUC0-48hr of 6-B-Naloxol Plasma Concentration
Description: AUC0-48hr of 6-B-Naloxol plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*pg/mL
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr*pg/mL | 1655.48 (667.02) | 5065.33 (3358.14)

34. Primary Outcome: AUC0-t of 6-B-Naloxol Plasma Concentration
Description: AUC0-t of 6-B-Naloxol plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*pg/mL
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr*pg/mL | 1373.11 (779.63) | 5049.62 (3374.52)

35. Primary Outcome: AUC_%Extrap of 6-B-Naloxol Plasma Concentration
Description: AUC_%Extrap of 6-B-Naloxol plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: (%)
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
(%) | 21.24 (15.98) | 33.37 (15.60)

36. Primary Outcome: AUCinf of 6-B-Naloxol Plasma Concentration
Description: AUCinf of 6-B-Naloxol plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: hr*pg/mL
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 0
hr*pg/mL | 1828.39 (878.66) |

37. Primary Outcome: Cmax of 6-B-Naloxol Plasma Concentration
Description: Cmax of 6-B-Naloxol plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
pg/mL | 85.18 (47.25) | 269.53 (189.50)

38. Primary Outcome: Lambda_z of 6-B-Naloxol Plasma Concentration
Description: Lambda_z of 6-B-Naloxol plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 0
1/hr | 0.07 (0.02) |

39. Primary Outcome: T1/2 of 6-B-Naloxol Plasma Concentration
Description: T1/2 of 6-B-Naloxol plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 0
hr | 9.78 (2.20) |

40. Primary Outcome: Tmax of 6-B-Naloxol Plasma Concentration
Description: Tmax of 6-B-Naloxol plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Median (Full Range); unit: hr
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr | 6.50 [0.50 to 14.00] | 1.75 [0.50 to 12.00]

41. Primary Outcome: AUC0-48hr of NLLG Plasma Concentration
Description: AUC0-48hr of NLLG plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*pg/mL
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr*pg/mL | 57735.72 (24399.37) | 209514.4 (104345.5)

42. Primary Outcome: AUC0-t of NLLG Plasma Concentration
Description: AUC0-t of NLLG plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*pg/mL
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr*pg/mL | 57737.49 (24400.80) | 209514.4 (104345.5)

43. Primary Outcome: AUC_%Extrap of NLLG Plasma Concentration
Description: AUC_%Extrap of NLLG plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: (%)
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
(%) | 13.13 (14.09) | 20.07 (9.23)

44. Primary Outcome: AUCinf of NLLG Plasma Concentration
Description: AUCinf of NLLG plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: hr*pg/mL
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 0
hr*pg/mL | 62953.71 (26257.03) |

45. Primary Outcome: Cmax of NLLG Plasma Concentration
Description: Cmax of NLLG plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
pg/mL | 3442.63 (1800.17) | 11372.74 (5426.77)

46. Primary Outcome: Lambda_z of NLLG Plasma Concentration
Description: Lambda_z of NLLG plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 0
1/hr | 0.07 (0.02) |

47. Primary Outcome: T1/2 of NLLG Plasma Concentration
Description: T1/2 of NLLG plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 0
hr | 11.32 (4.26) |

48. Primary Outcome: Tmax of NLLG Plasma Concentration
Description: Tmax of NLLG plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Median (Full Range); unit: hr
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr | 11.00 [0.50 to 14.00] | 1.50 [0.50 to 7.00]

49. Primary Outcome: AUC0-48hr of NLXG Plasma Concentration
Description: AUC0-48hr of NLXG plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*pg/mL
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr*pg/mL | 78725.81 (28285.24) | 320734.4 (113332.8)

50. Primary Outcome: AUC0-t of NLXG Plasma Concentration
Description: AUC0-t of NLXG plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*pg/mL
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr*pg/mL | 77976.24 (28477.82) | 320734.4 (113332.8)

51. Primary Outcome: AUC_%Extrap of NLXG Plasma Concentration
Description: AUC_%Extrap of NLXG plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: (%)
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
(%) | 1.56 (1.05) | 1.86 (1.39)

52. Primary Outcome: AUCinf of NLXG Plasma Concentration
Description: AUCinf of NLXG plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*pg/mL
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr*pg/mL | 79025.78 (28389.19) | 326907.3 (115103.6)

53. Primary Outcome: Cmax of NLXG Plasma Concentration
Description: Cmax of NLXG plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
pg/mL | 11488.62 (2493.48) | 45789.83 (10576.00)

54. Primary Outcome: Lambda_z of NLXG Plasma Concentration
Description: Lambda_z of NLXG plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
1/hr | 0.14 (0.03) | 0.09 (0.03)

55. Primary Outcome: T1/2 of NLXG Plasma Concentration
Description: T1/2 of NLXG plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr | 5.28 (1.35) | 8.40 (2.43)

56. Primary Outcome: Tmax of NLXG Plasma Concentration
Description: Tmax of NLXG plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Median (Full Range); unit: hr
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr | 1.01 [0.50 to 8.00] | 1.25 [0.50 to 3.00]

57. Primary Outcome: AUC0-48hr of Naloxone Plasma Concentration
Description: AUC0-48hr of Naloxone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*pg/mL
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr*pg/mL | 281.91 (122.61) | 650.42 (222.44)

58. Primary Outcome: AUC0-t of Naloxone Plasma Concentration
Description: AUC0-t of Naloxone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*pg/mL
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr*pg/mL | 136.17 (92.95) | 443.88 (252.95)

59. Primary Outcome: AUC_%Extrap of Naloxone Plasma Concentration
Description: AUC_%Extrap of Naloxone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: (%)
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
(%) | 47.82 (20.95) | 44.94 (26.95)

60. Primary Outcome: AUCinf of Naloxone Plasma Concentration
Description: AUCinf of Naloxone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Population: as for outcome 28
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 0 | 0

61. Primary Outcome: Cmax of Naloxone Plasma Concentration
Description: Cmax of Naloxone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
pg/mL | 33.21 (24.62) | 45.10 (21.03)

62. Primary Outcome: Lambda_z of Naloxone Plasma Concentration
Description: Lambda_z of Naloxone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Population: as for outcome 28
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 0 | 0

63. Primary Outcome: T1/2 of Naloxone Plasma Concentration
Description: T1/2 of Naloxone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Population: as for outcome 28
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 0 | 0

64. Primary Outcome: Tmax of Naloxone Plasma Concentration
Description: Tmax of Naloxone plasma concentration. Plasma concentrations of OXN 5/2.5 mg and OXN 20/10mg Will be Analyzed.
Time Frame: as for outcome 3
Measure: Median (Full Range); unit: hr
Arm/Group | OXN Prolonged Release Tablet 5/2.5mg | OXN Prolonged Release Tablet 20/10mg
Number analyzed (Participants) | 12 | 12
hr | 8.00 [5.00 to 14.00] | 1.00 [0.50 to 8.00]

ADVERSE EVENTS:
Time Frame: Events will be recorded from the point at which the Informed Consent is signed until 7(+3) days after the subject leaves the study.
Arm/Group | OXN PR Tablet 5/2.5 mg | OXN PR Tablet 20/10 mg
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/17
Other Adverse Events (participants affected / at risk) | 9/13 | 13/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OXN PR Tablet 5/2.5 mg (N=13) | OXN PR Tablet 20/10 mg (N=17)
upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OXN PR Tablet 5/2.5 mg (N=13) | OXN PR Tablet 20/10 mg (N=17)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Elevated aminotransferase (Investigations) | 1 (1) | 0 (0)
Sleepiness (Nervous system disorders) | 4 (4) | 6 (6)
headache (Nervous system disorders) | 3 (3) | 1 (1)
dizziness (Nervous system disorders) | 2 (2) | 5 (5)
vertigo (Nervous system disorders) | 0 (0) | 1 (1)
Imbalance of autonomic nervous system (Nervous system disorders) | 0 (0) | 1 (1)
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
dry pharynx (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
flushing (General disorders) | 0 (0) | 1 (1)
fatigue (General disorders) | 0 (0) | 1 (1)
cold sweat (General disorders) | 0 (0) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 5 (5)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
vomit (Gastrointestinal disorders) | 1 (1) | 5 (5)
Difficult defecation (Gastrointestinal disorders) | 3 (3) | 3 (3)
toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
palpitation (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2014-09-25): https://cdn.clinicaltrials.gov/large-docs/75/NCT02880475/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT02880475/SAP_001.pdf